CLINICAL TRIAL: NCT02373358
Title: A Mixed Methods Evaluation of Effectiveness of a Group Yoga Intervention as an Adjunctive Trauma Therapy for Adolescent Girls
Brief Title: Evaluation of Effectiveness of a Group Yoga Intervention as Trauma Therapy for Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 700871-1
Record Dates: First submitted 2015-02-09; First posted 2015-02-27 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: PTSD
Keywords: Complex trauma; Yoga
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Group yoga intervention (Experimental): Participants will participate in 6 90-minute yoga groups designed to promote themes related to trauma recovery (safety & boundaries, strength & power, assertiveness, intuition, trust, & community) using mindfulness, breath work, and physical yoga poses.
  Interventions: Behavioral: Group yoga intervention

INTERVENTIONS:
Behavioral: Group yoga intervention — Participants will participate in 6 90-minute yoga groups designed to promote themes related to trauma recovery (safety & boundaries, strength & power, assertiveness, intuition, trust, & community) using mindfulness, breath work, and physical yoga poses.

SUMMARY:
Neuroscience evidence indicates that trauma is stored in the body, that trauma impairs the language centers found in the brain, and that emotion centers in the brain tend to override cognitive centers in the brain following trauma. Most evidence-based models to date to treat trauma using cognitive therapy, which does not fully resolve symptoms, particularly in the case of complex trauma. This evidence has led to researchers to call for alternative, body-oriented treatments that target trauma from the lowest levels of regulation up to higher levels of regulation in the brain. Yoga has been proposed as one such intervention. Recent research has investigated the benefits of yoga to treatment adult females who have experienced PTSD, but only anecdotal, descriptive, and qualitative data is available for studies of yoga with adolescents. This mixed methods study seeks to generate quantitative data demonstrating whether or not the 6-week group yoga intervention leads to decreases in general mental health and trauma-specific symptoms and qualitative data regarding the components of the intervention the participants found both helpful and unhelpful.

DETAILED DESCRIPTION:
A mixed methods design was chosen for this study due to the study representing a new stream of literature, and a desire to capture the fullest picture possible regarding the participants' response to the intervention. The purpose of this mixed methods study is to generate quantitative data that demonstrates a decrease in trauma and general mental health symptoms following a yoga psychotherapy intervention for trauma, and to collect qualitative data during the group process and following the group that provides a picture of the mechanisms that allow the intervention to be effective. Broad Hypotheses: Quantitatively, there will be significant differences in total number of mental health symptoms and trauma-related symptoms experienced from pretest to posttest. Qualitative data will demonstrate the benefits from the yoga postures and experiences of relaxing breath work the youth experienced during the yoga group.

Trauma is a prevalent experience in our society, with between 50-76% of individuals experiencing a traumatic event with the potential to cause Posttraumatic Stress Disorder. The current standard of care in trauma treatment largely involves cognitive interventions, but neuroscience evidence demonstrates reasons for their limited effectiveness and a need to help traumatized individuals regulate the brain from the lowest levels up. Neuroscience research indicates the brains of individuals who have experienced trauma are less able to use cognitive centers to suppress emotional fear responses, and language centers in the brain experience deactivation during traumatic events. Indeed, 33% of individuals who develop PTSD fail to recover fully, which leads to ongoing mental health difficulties, impaired interpersonal relationships, substance abuse, physical health problems, and sexual problems.

Yoga has been proposed as a somatic, bottom-up intervention that allows the individual to regulate from the lowest level of the brain to higher levels of the brain by working with the body and mindful experience in the present moment. Existing investigation of yoga as a psychotherapeutic intervention is preliminary, but promising. van der Kolk and colleagues conducted a preliminary randomized controlled study and found that over 50% of individuals who participated in the yoga group no longer met criteria for Posttraumatic Stress Disorder following the group. Carmody and Baer found that yoga-based interventions in Mindfulness-Based Stress Reduction impacted the widest range of symptoms (compared to body scans and seated meditation). No quantitative investigations of trauma-related yoga treatment for adolescents have been conducted, other than one dissertation with juvenile sex offenders. Existing yoga psychotherapy research on youth who have experienced trauma has been qualitative in nature with case studies and limited samples.

Additional study of yoga as an intervention for traumatized adolescents is needed both quantitatively and qualitatively. One model of group yoga as adjunctive treatment for trauma has been identified in the literature, but it has only been described anecdotally and with limited qualitative data. Thus, the aim of the current study is to use the model created for the Healing Childhood Sexual Abuse with Yoga curriculum with a wider sample of adolescents across types of trauma (emotional, physical, & sexual abuse & neglect) in the United States and Canada to generalize the curriculum and generate qualitative and quantitative data regarding its effectiveness and the perceived mechanisms that contribute to success. Additional qualitative research would be beneficial to describe the themes and cases across a full sample of participants in such a group. Current research has been observational, case studies, or limited qualitative questionnaires at the end of the group, but this study proposes to collect qualitative data at each group yoga session regarding the experience. In addition, follow-up interviews are also proposed to ask more detailed questions about the participants' experiences.

Participants will be referred from within the agencies providing the groups, and therapists will complete an internal referral form providing minimal demographic data with the referral. Participants will be contacted by the respective group leaders at the phone numbers listed on the referrals forms. Prior to the beginning of the initial group, the group leaders will meet with prospective clients to interview them for appropriateness for the group, obtain informed consent and assent, and allow them to complete the pretest measures. In addition to obtaining informed consent for the research process, the group leader will explain the physical nature of the yoga group, and the group leader will obtain waivers from parents for the youth to participate in the physical activity involved in the group. Copies of consent and assent forms will be provided to participants and parents.

During each group, participants will complete the Yoga Experience Form at each session. Posttests will be completed at the end of the sixth group meeting. They will include all the pretest questionnaires, as well as the Therapeutic Factors Inventory- Cohesiveness Scale and the Working Alliance Inventory-Short Form- Bond Scale. After the final group, pretest, within, and posttest data will be coded and analyzed to determine the questions to be utilized for the follow-up interviews. Two participants from each group at McMaster Children's Hospital will be asked to complete a follow-up interview with the investigator that will be approximately 30 minutes in length. Participants will be selected with well defined symptom improvement and poor response to the intervention. The follow-up interviews will be audio recorded. Willingness to be audio recorded is necessary for participation in the follow-up interviews, but not for participation in the larger group. The time commitment for the treatment group is 540 minutes. This study does not involve additional post-treatment follow-up, aside from clients who volunteer to participate in the follow-up interviews.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between the ages of 11 and 18
* Current participation in outpatient treatment at the Denver Children's Advocacy Center or McMaster Children's Hospital (Regional and Outpatient Services).
* History of complex trauma with clinical or subclinical PTSD symptoms

Exclusion Criteria:

* Non-English-speaking individuals.
* Currently suicidal, homicidal, or psychotic
* Significant substance use (daily or greater use of marijuana or weekly or greater use of other non-prescription/illegal drugs)

Ages: 11 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in general mental health symptoms at 6 weeks | Entry & at 6 weeks
  The Youth Outcomes Questionnaire-Self Report (YOQ-SR) is used to evaluate treatment outcomes based on global symptom reduction (Wells, Burlingame, & Lambert, 2003). The YOQ is very sensitive to change, and individuals are asked to report on their symptoms within the last seven days. The 64-item questionnaire produces a total score of -16 to 240 (due to negative scores being awarded for reverse-scored items, a negative score is possible). Symptoms are rated on a 5-point Likert scale from Never or Almost Never to Almost Always or Always. Questions include, "I want to be alone more than others my same age," "My emotions are strong and change quickly," "I am calm," and "I don't forgive myself for things I've done wrong." The YOQ-SR was chosen due to its ease of use, brief administration time, sensitivity to change, and previous data supporting strong reliability and validity (Wells, Burlingame, & Lambert, 2003).
Change from baseline in PTSD symptoms | Entry & at 6 weeks
  The Child PTSD Symptom Scale (CPSS) assesses PTSD symptom severity in children 8-18 based on Diagnostic and Statistical Manual or Mental Disorders, 4th edition diagnostic criteria (Foa, Johnson, Feeny, & Treadwell, 2001). It includes 17 items that map onto diagnostic criteria, & 7 items assessing functional impairment caused by the PTSD symptoms. It can be completed in 10 minutes. Part one of the questionnaire involves a 4-point Likert-like scale (from 0=not at all or only at one time to 3=5 or more times a week/almost always), and part two involves dichotomous questions. The measure yields a total score from 0 to 51 with a clinical cutoff of 15, and also provides three subscale scores for re-experiencing, avoidance, and hyperarousal. The measure is relatively time-sensitive, asking respondents to indicate how many times a problem has bothered her in the last two weeks.

SECONDARY OUTCOMES:
Change from baseline in trauma-related beliefs | Entry & and at 6 weeks
  The author developed an affirmation questionnaire corresponding to the affirmations/mantras used in each group. For example, affirmations included "I believe that I have the right to be safe," "I can tell others 'no' when they intrude in my personal space," and "I feel that I am strong." In addition, two general questions were included that asked about the client's ability to regulate her emotions and having skills that help her cope with her trauma. Responses are scored on a 5-point Likert scale with scores ranging from 1= strongly disagree to 5= strongly agree. Total scores for this questionnaire range from 10 to 50.
Therapeutic Factors Inventory- Cohesiveness Scale | After 6 weeks of intervention
  This measure was chosen to address potential effects of group cohesion that contributed to the study outcomes to control for this effect, and will be given after the group intervention. The nine-item Cohesiveness scale measures socio-emotional aspects of group cohesion (MacNair-Semands & Lese, 2000), drawing on Yalom's (1995) therapeutic factors. Responses are rated on a 7-point Likert-like scale from strongly disagree=1 to strongly agree=7. Items include "I feel accepted by the group," "I feel a sense of belonging in the group," and "We trust each other in my group." Previous test-retest reliability of 0.93 was reported, as well as a previous a level of 0.90 (MacNair-Semands & Lese, 2000).
Working Alliance Inventory- Short Form- Bond Scale | After 6 weeks of intervention
  The Working Alliance Inventory - Short Form (WAI-S) (Tracey & Kokotovic, 1989) is a 12-item 5-point Likert measure derived from the original 36-item version (Horvath & Greenberg, 1989) that assesses the three dimensions of agreement on pertinent therapeutic tasks (Tasks), agreement on therapeutic goals (Goals), and development of affective bonds between client and therapist (Bond). Tracey and Kokotovic (1989) reported evidence supporting the construct validity of the WAI - Short Form, as well as high internal consistency estimates from .83 to .98 for its three factors. This study is using the 4-item bonds scale in order to control for the effects of the therapeutic alliance on the group. Items include "I believe ___ likes me," and "I feel that ____ appreciates me."
Interviews to assess benefits and limitations of the group yoga intervention following group | After 6 weeks of intervention
  Follow-up qualitative interviews will be conducted with a subset of group participants. An even number of participants will be selected from each group, and attempts will be made to balance the number of participants with PTSD diagnoses and with subclinical symptoms and those who benefited from the group and did not. Questions include: 1. In what ways do you think yoga contributed to the experience of this group? 2. In what ways do you think being in a group affected this experience? 3. Would you do this group again if offered? Why or why not? 4. What were some important things/the most important thing you learned about yourself from these sessions? 5. What wasn't helpful for you about these sessions? 6. Were any of the themes easier or more difficult to relate to than others?
Weekly Yoga Experiences Form | Weekly for 6 weeks
  During each session, clients will fill out a Yoga Experiences Form rating their levels of calmness versus distress on a scale of 1 to 10 prior to the group and then following the group, as well as commenting on content of the group that they found helpful and difficult, that came into their awareness, and that they want to practice again.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia McRae, PhD, Study Chair — University of Denver; Paulo Pires, PhD, Study Director — Hamilton Health Sciences Corporation
Locations (2):
- Denver Children's Advocacy Center, Denver, Colorado, United States
- Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Carmody J, Baer RA. Relationships between mindfulness practice and levels of mindfulness, medical and psychological symptoms and well-being in a mindfulness-based stress reduction program. J Behav Med. 2008 Feb;31(1):23-33. doi: 10.1007/s10865-007-9130-7. Epub 2007 Sep 25. PMID 17899351
- [Background] Copeland WE, Keeler G, Angold A, Costello EJ. Traumatic events and posttraumatic stress in childhood. Arch Gen Psychiatry. 2007 May;64(5):577-84. doi: 10.1001/archpsyc.64.5.577. PMID 17485609
- [Background] Dale, L. P., Carroll, L. E., Galen, G. C., Schein, R., Bliss, A., Mattison, A. M., & Neace, W. P. (2011). Yoga practice may buffer the deleterious effects of abuse on women's self-concept and dysfunctional coping. Journal of Aggression, Maltreatment, & Trauma, 20, 89-101.
- [Background] D'Andrea W, Ford J, Stolbach B, Spinazzola J, van der Kolk BA. Understanding interpersonal trauma in children: why we need a developmentally appropriate trauma diagnosis. Am J Orthopsychiatry. 2012 Apr;82(2):187-200. doi: 10.1111/j.1939-0025.2012.01154.x. PMID 22506521
- [Background] Dick AM, Niles BL, Street AE, DiMartino DM, Mitchell KS. Examining mechanisms of change in a yoga intervention for women: the influence of mindfulness, psychological flexibility, and emotion regulation on PTSD symptoms. J Clin Psychol. 2014 Dec;70(12):1170-82. doi: 10.1002/jclp.22104. Epub 2014 May 28. PMID 24888209
- [Background] Emerson, D., Sharma, R., Chaudhry, S. & Turner, J. (2009). Trauma-sensitive yoga: Principles, practice, and research. International Journal of Yoga Therapy, 19, 123-128.
- [Background] Foa EB, Johnson KM, Feeny NC, Treadwell KR. The child PTSD Symptom Scale: a preliminary examination of its psychometric properties. J Clin Child Psychol. 2001 Sep;30(3):376-84. doi: 10.1207/S15374424JCCP3003_9. PMID 11501254
- [Background] Koenigs M, Grafman J. Posttraumatic stress disorder: the role of medial prefrontal cortex and amygdala. Neuroscientist. 2009 Oct;15(5):540-8. doi: 10.1177/1073858409333072. Epub 2009 Apr 9. PMID 19359671
- [Background] Horvath, A. O., Greenberg, L. S. (1989). Development and validation of the Working Alliance Inventory. Journal of Counseling Psychology, 36(2), 223-233.
- [Background] Lilly, M., & Hedlund, J. (2010). Yoga therapy in practice: Healing childhood sexual abuse with yoga. International Journal of Yoga Therapy, 20, 120-130.
- [Background] MacNair-Semands, R. R., & Lese, K. P. (2000). Interpersonal problems and the perception of therapeutic factors in group therapy. Small Group Research, 31(2), 158-174.
- [Background] McLaughlin KA, Koenen KC, Hill ED, Petukhova M, Sampson NA, Zaslavsky AM, Kessler RC. Trauma exposure and posttraumatic stress disorder in a national sample of adolescents. J Am Acad Child Adolesc Psychiatry. 2013 Aug;52(8):815-830.e14. doi: 10.1016/j.jaac.2013.05.011. Epub 2013 Jun 25. PMID 23880492
- [Background] McRae, K., Ochsner, K. N., & Gross, J. J. (2011). The reason in passion: A social cognitive neuroscience approach to emotion regulation (Chapter 10). In Handbook of Self-Regulation, Second Edition: Research, Theory, and Applications. New York: The Guilford Press.
- [Background] Michalsen A, Jeitler M, Brunnhuber S, Ludtke R, Bussing A, Musial F, Dobos G, Kessler C. Iyengar yoga for distressed women: a 3-armed randomized controlled trial. Evid Based Complement Alternat Med. 2012;2012:408727. doi: 10.1155/2012/408727. Epub 2012 Sep 25. PMID 23049608
- [Background] Mitchell KS, Dick AM, DiMartino DM, Smith BN, Niles B, Koenen KC, Street A. A pilot study of a randomized controlled trial of yoga as an intervention for PTSD symptoms in women. J Trauma Stress. 2014 Apr;27(2):121-8. doi: 10.1002/jts.21903. Epub 2014 Mar 25. PMID 24668767
- [Background] Neumann, D. A., Houskamp, B. M., Pollock, V. E., & Briere, J. (1996). The long-term sequelae of childhood sexual abuse in women: A meta-analytic review. Child Maltreatment, 1(1), 6-16.
- [Background] Pelcovitz D, Kaplan S, Goldenberg B, Mandel F, Lehane J, Guarrera J. Post-traumatic stress disorder in physically abused adolescents. J Am Acad Child Adolesc Psychiatry. 1994 Mar-Apr;33(3):305-12. doi: 10.1097/00004583-199403000-00002. PMID 8169174
- [Background] Perry, B. D. (2009). Examining child maltreatment through a neurodevelopmental lens: Clinical applications of the Neurosequential Model of Therapeutics. Journal of Loss & Trauma, 14, 240-255.
- [Background] Tracey, T. J., & Kokotovic, A. M. (1989). Factor structure of the Working Alliance Inventory. Psychological Assessment, 1, 207- 210.
- [Background] Van Ameringen M, Mancini C, Patterson B, Boyle MH. Post-traumatic stress disorder in Canada. CNS Neurosci Ther. 2008 Fall;14(3):171-81. doi: 10.1111/j.1755-5949.2008.00049.x. PMID 18801110
- [Background] van der Kolk, B. A. (2005). Developmental trauma disorder. Psychiatric Annals, 35(5), 401-408.
- [Background] van der Kolk BA. Clinical implications of neuroscience research in PTSD. Ann N Y Acad Sci. 2006 Jul;1071:277-93. doi: 10.1196/annals.1364.022. PMID 16891578
- [Background] van der Kolk BA, Stone L, West J, Rhodes A, Emerson D, Suvak M, Spinazzola J. Yoga as an adjunctive treatment for posttraumatic stress disorder: a randomized controlled trial. J Clin Psychiatry. 2014 Jun;75(6):e559-65. doi: 10.4088/JCP.13m08561. PMID 25004196
- [Background] Wells, M. G., Burlingame, G. M., & Lambert, P. M. (2003). Y-OQ-SR2.0: Administration & Scoring Manual. Salt Lake City, UT: OQ Measures, LLC.
- [Background] Yalom, I. D. (1995). The Theory and Practice of Group Psychotherapy. New York: Basic Books.